CLINICAL TRIAL: NCT05567263
Title: Post-operative Sensitivity and Clinical Performance of a Self-adhesive Restorative Material in Posterior Restorations.
Brief Title: Post-operative Sensitivity of a Self-adhesive Restorative Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ghada Maghaireh, Principal Investigator, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210419
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Dental Restorations, Permanent
Keywords: Composite, self-adhesive, sensetivity

STUDY DESIGN:
Intervention Model Description: The design of study will be a split-mouth randomized clinical trial with two study groups.
Who Masked: Participant
Masking Description: All participants will be informed about the nature and objectives of the study; however, they will not be informed what material they would receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulk- Fill (Active Comparator): Restorative procedure of the teeth will be performed using Filtek-Bulk Fill Posterior Restorative, Bulk-fill resin composite, (3M, ESPE) following application of an etch-and-rinse single bottle adhesive (3M, ESPE).
  Interventions: Procedure: Bulk-fill resin composite, (3M, ESPE)
- Surefill One (Experimental): Restorative procedure of the teeth will be performed using Surefil one™ Self-Adhesive Composite Hybrid (Dentsply, Sirona),
  Interventions: Procedure: Surefil one™ Self-Adhesive Composite Hybrid

INTERVENTIONS:
Procedure: Bulk-fill resin composite, (3M, ESPE) — Teeth will be restored with Bulk-fill resin composite, (3M, ESPE)
  Arms: Bulk- Fill
Procedure: Surefil one™ Self-Adhesive Composite Hybrid — teeth will be restored with Surefil one™ Self-Adhesive Composite Hybrid
  Arms: Surefill One

SUMMARY:
Adhesively restoring teeth using a resin-based composite and a modern dental adhesive is now considered a reliable, predictable, and durable procedure. However, adhering resin-based composite in conditions of suboptimal field control or complex cavity configurations remains challenging. In addition, the continuing discussions on the clinical use of dental amalgam and the feasibility of a phase out of the use of dental amalgam in the long term has become a central concern for restorative dentistry and has led to strong efforts to develop a substitute material for amalgam. With the goal of clinically shorter application times and lower technique sensitivity, the development of an advanced self-adhesive restorative tooth-colored restorative materials (ASAR) that no longer need pre-treatment with a separate adhesive have been under investigation. The aim of this study is to assess the post-operative sensitivity following restoration of teeth using a self-adhesive tooth-colored restorative material and to assess its clinical performance in comparison with conventional resin-based composite in posterior restorations

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years' old
* Teeth are vital
* Teeth are periodontal healthy
* Tooth to be restored in normal occlusion with natural antagonist and adjacent teeth
* Patient did not receive orthodontic treatment
* Good level of oral hygiene.

Exclusion Criteria:

* Non-vital or endodontically treated teeth
* (Profound, chronic) periodontitis
* Deep carious defects (close to pulp, < 1mm distance)
* Heavy occlusal contacts or history of bruxism
* Poor oral hygiene
* Sustained dentin hypersensitivity
* Taking anti-inflammatory, analgesic, or psychotropic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The post-operative sensitivity. | One month after the treatment.
  For the evaluation of post-operative sensitivity, participants will be asked to record whether they experienced sensitivity using a 0-4 numerical rating scale (0 = none, 1 = mild, 2 = moderate, 3 = considerable, and 4 = severe). The patients will be asked to fill in the pain scale forms 24 hours after the restorative procedure and daily up to seven days, and at 2 weeks and 1 month intervals.

SECONDARY OUTCOMES:
Clinical performance of the restorations | 6 months and 1 year after the treatment.
  All restorations will be evaluated at 6 months and 1-year post-restoration using the United States Public Health Service, USPHS criteria using the Alpha, Bravo and Charlie scale to evaluate the following parameters: retention, color match, marginal discoloration, secondary caries, anatomical form, marginal adaptation, and surface roughness.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Maghaireh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maghaireh GA, Albashaireh ZS, Allouz HA. Postoperative sensitivity in posterior restorations restored with self-adhesive and conventional bulk-fill resin composites: A randomized clinical split-mouth trial. J Dent. 2023 Oct;137:104655. doi: 10.1016/j.jdent.2023.104655. Epub 2023 Aug 9. PMID 37562757